CLINICAL TRIAL: NCT00043901
Title: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Evaluation of Lamotrigine Adjunctive Therapy in Subjects Wtih Primary Generalized Tonic-Clonic Seizures
Brief Title: Treatment Of Primary Generalized Tonic-Clonic Seizures With An Investigational New Drug
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAM40097
Record Dates: First submitted 2002-08-14; First posted 2002-08-16 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Epilepsy, Tonic-Clonic
Keywords: PGTC; Lamotrigine; epilepsy; seizures; primary generalized tonic-clonic
MeSH Terms: conditions — Epilepsy, Tonic-Clonic; Epilepsy; Seizures | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of an investigational new drug for supplemental therapy in subjects with primary generalized tonic-clonic (PGTC) seizures.

ELIGIBILITY:
INCLUSION CRITERIA:

* Weigh at least 13kg.
* Have a confident diagnosis of epilepsy with primary generalized tonic-clonic (PGTC) seizures with or without other generalized seizure types.
* Currently being treated with an antiepileptic drug(s) (AED).
* Benzodiazepines are allowed with some frequency restrictions.
* Vagus nerve stimulation is allowed if in place for at least 6 months prior to starting the study with no changes to the settings having occured during the month immediately prior to starting the study, and if no changes will occur during all phases of the study.
* History of primary generalized tonic-clonic seizures with no focal onset.
* Have at least 1 primary generalized tonic-clonic (PGTC) seizure during the 8 consecutive weeks prior to the baseline period of the study.
* Have at least 3 PGTC seizures occur anytime during the 8-week baseline phase of the study.
* Females must agree to acceptable form of birth control.

EXCLUSION CRITERIA:

* A history of partial seizures or interictal expression of partial seizures as evidenced by electroencephalogram.
* Have Lennox-Gastaut syndrome.
* Currently using or has previously used the drug being studied.
* Is abusing alcohol and/or other substance(s).
* Has taken an investigational drug during the 30 days prior to the study or plans to take an investigational drug anytime during the study.
* Is receiving chronic (long-term) treatment with any medication that could influence seizure control.
* Follows the ketogenic diet.
* Is planning surgery to control seizures during the study.
* Is suffering from acute or progressive neurological disease, severe psychiatric disease, or severe mental abnormality.
* Has any clinically significant heart, kidney, or liver condition, or a condition that affects how drugs are absorbed, distributed, metabolized, or removed from the body.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2000-12-01; Primary Completion 2003-11-01 (Actual); Study Completion 2005-03-01 (Actual)

PRIMARY OUTCOMES:
% change from Baseline in average monthly PGTC seizure frequency

SECONDARY OUTCOMES:
Proportion of subjects with >/= 25%, 50%, 75% or 100% reduction in PGTC seizures %change from Baseline in average monthly seizure frequency.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (79):
- United States (74):
  - GSK Investigational Site, Alabaster, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Northport, Alabama
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Gainsville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Crestview Hills, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Newton, Massachusetts
  - GSK Investigational Site, Sharon, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Saint Cloud, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Medford, New Jersey
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Mount Vernon, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Danville, Pennsylvania
  - GSK Investigational Site, Natrona Heights, Pennsylvania
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Bennington, Vermont
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (2):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Capital Federal
- Chile (2):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, San Isidro, Lima region, Peru

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Biton V, Sackellares JC, Vuong A, Hammer AE, Barrett PS, Messenheimer JA. Double-blind, placebo-controlled study of lamotrigine in primary generalized tonic-clonic seizures. Neurology. 2005 Dec 13;65(11):1737-43. doi: 10.1212/01.wnl.0000187118.19221.e4. PMID 16344515
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: LAM40097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LAM40097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM40097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM40097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM40097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM40097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LAM40097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register